CLINICAL TRIAL: NCT00005928
Title: Effects of Angiotensin Converting Enzyme Inhibitor Therapy on Vascular Inflammation and Compliance
Brief Title: Effects of Angiotensin-Converting Enzyme Inhibitor (Ramipril) Therapy on Blood Vessel Inflammation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000162; 00-H-0162
Record Dates: First submitted 2000-06-28; First posted 2000-06-29 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-02

CONDITIONS: Atherosclerosis; Coronary Disease; Vasculitis
Keywords: ACE Inhibitor; Vascular Inflammation; Vascular Compliance; Cell Adhesion Molecules; Coronary Artery Disease
MeSH Terms: conditions — Atherosclerosis; Coronary Disease; Vasculitis; Coronary Artery Disease | interventions — Ramipril

INTERVENTIONS:
Drug: Ramipril

SUMMARY:
This study will determine the effects of angiotensin-converting enzyme (ACE) inhibitor (trade name Ramipril) therapy on inflammation and stiffness of artery walls. These are two risk factors for developing atherosclerosis-deposits of fatty substances called plaques that can block the blood vessel, causing a heart attack or stroke. Studies of patients with coronary artery disease suggest that ACE inhibitor therapy reduces the risk of heart attack and heart failure. This study will examine the effects of this treatment on the artery walls and on levels of substances in the blood that indicate blood vessel inflammation.

Patients between 40 and 75 years old with coronary artery disease caused by atherosclerosis may be eligible for this study. Candidates will be screened with a medical history, cardiovascular (heart and blood vessel) examination, electrocardiogram and blood tests. Those enrolled will be randomly assigned to take either an ACE inhibitor pill or a placebo (look-alike pill with no medicine) once a day for 3 months. No pills will be taken for the next month, and then participants will take the alternate pill for the next 3 months. That is, those who took ACE inhibitor for the first 3-month period will take placebo for the second 3-month period and vice versa. Blood pressures will be taken at the NIH Clinical Center or by the patient's physician at the end of the first and second weeks of the study. At the end of 3 weeks, patients will return to the Clinical Center for a blood draw of 6 cc (1/2 teaspoon) to assess kidney function. In addition, at the end of each 3-month study period, patients will undergo the following procedures at the Clinical Center:

1. Fasting blood draw of 60 cc (2 ounces) to measure electrolytes (e.g., sodium and potassium) and blood markers for inflammation
2. Ultrasound (use of sound waves to create pictures) study of the carotid arteries (arteries in the neck leading to the brain)-An ultrasound probe is applied gently on the neck, and ultrasound pictures of the right and left carotid arteries are recorded on tape. Heart activity and blood pressure are monitored during the procedure with an electrocardiogram and blood pressure cuff.
3. Magnetic resonance imaging (MRI) of the carotid arteries-The patient lies on a table in a narrow cylinder (the MRI machine) containing a magnetic field. A flexible padded sensor called a MRI coil is placed over the neck area. Earplugs are placed in the ear to muffle the loud thumping sounds the machine makes when the magnetic fields are switched. During the second half of the exam, a contrast agent (gadolinium) is injected through an intravenous catheter (flexible tube placed in a vein) to brighten the images. The heart is monitored during the procedure with an electrocardiogram.

DETAILED DESCRIPTION:
Vascular inflammation plays a major role in the progression and clinical expression of atherosclerosis and may contribute to stiffening of arteries that increases the risk of myocardial infarction and stroke. Therapies that reduce vascular inflammation may reduce cardiovascular events. Angiotensin converting enzyme (ACE) inhibitor therapy reduces cardiovascular events in patients with coronary artery disease (CAD), potentially by reducing vascular oxidant stress and activation of genes that encode protein mediators of inflammation. However, we found that ACE inhibitor therapy in patients with CAD had no overall significant effect on serum levels of cell adhesion molecules VCAM-1, ICAM-1, and E-selectin (surrogate markers of vascular inflammation), although some patients showed a reduction in levels, suggesting either that these surrogate markers of vascular inflammation may not accurately reflect reduction in vascular inflammation, or that only a subset of patients have biological responses that might reduce their cardiovascular risk. The purposes of this protocol are to determine 1) the effect of ACE inhibitor therapy on vascular inflammation in patients with coronary artery disease as assessed by MRI of the carotid arteries, and 2) whether serum markers of inflammation correlate with reduced vascular inflammation and thus may be suitable surrogates for determining success of ACE inhibitor therapy.

ELIGIBILITY:
All volunteer subjects must be between 40 and 75 years of age with documented CAD, and must have provided informed, written consent for participation in this study.

Ability to comprehend or willingness to sign the consent form.

No pregnant women or women with child-bearing potential not on effective contraception.

No ACE inhibitor therapy within 6 months.

No renal insufficiency (creatinine greater than 2.0 mg/dl).

Blood pressure must not be higher than 140/90 on current medical therapy.

No claustrophobia.

No history of involuntary motion disorder.

Specific MRI exclusion criteria (i.e. pacemaker, cochlear implants, AICD, internal infusion pump, metal implants or clips in field of view).

No systemic inflammatory disorder (e.g, rheumatoid arthritis, periarteritis nodosa, systemic lupus erythromatosus, temporal arteritis).

No need for chronic NSAID therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 2000-06; Study Completion 2002-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Liuzzo G, Biasucci LM, Gallimore JR, Grillo RL, Rebuzzi AG, Pepys MB, Maseri A. The prognostic value of C-reactive protein and serum amyloid a protein in severe unstable angina. N Engl J Med. 1994 Aug 18;331(7):417-24. doi: 10.1056/NEJM199408183310701. PMID 7880233
- [Background] Berliner JA, Navab M, Fogelman AM, Frank JS, Demer LL, Edwards PA, Watson AD, Lusis AJ. Atherosclerosis: basic mechanisms. Oxidation, inflammation, and genetics. Circulation. 1995 May 1;91(9):2488-96. doi: 10.1161/01.cir.91.9.2488. PMID 7729036
- [Background] Koh KK, Bui MN, Hathaway L, Csako G, Waclawiw MA, Panza JA, Cannon RO 3rd. Mechanism by which quinapril improves vascular function in coronary artery disease. Am J Cardiol. 1999 Feb 1;83(3):327-31. doi: 10.1016/s0002-9149(98)00862-5. PMID 10072217